CLINICAL TRIAL: NCT06197542
Title: Effects of Active Release Technique and Instrument Assisted Soft Tissue Mobilization in Patients With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/015
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Migraine Disorders
Keywords: Trigger points,; Active release Technique,; IATSM
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to the A group or B group after a baseline assessment with a lottery ticket and an opaque envelope containing the same number of folded papers labeled "Group A" or "Group B." Each participant took a piece of paper that identified their group and gave it to the researchers without seeing what was written. Participants were not notified which group was assigned to.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers who evaluated the participants were not informed of how the participants were grouped. Participants were informed that they would receive one of two different interventions without indicating which group should undergo trunk stability or conventional physiotherapy program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Technique (Experimental): Individuals in Group A will be subjected to Heat Therapy over the targeted muscles via hot pack for 5 minutes in every session along with passive stretching for 5 minutes Group A will receive Active release technique on targeted muscles. The participant was comfortably seated and rested the forehead on the forearms .To apply for the release, the active TrP was identified, and sustained and constant pressure was applied. For stretching of the SCM muscle, the patient performed contralateral lateral flexion and ipsilateral rotation of the head to achieve stretching, for trapezius the therapist performed lateral flexion of the neck.The treatment regimen will span over 3 weeks with a follow up frequency of 2 sessions per week.
  Interventions: Other: Active Release Technique
- Instrument Assisted Soft Tissue Mobilization (Experimental): Group A will be subjected to Heat Therapy for 5minutes along with Stretching for 5 minutes .Group B will be Subjected to IASTM using M2T blade for approximately 3 minutes per muscle. Lubricant was applied and the tool was cleaned with an alcohol pad.the tool was used to locate soft tissue restrictions in the muscles. Then, the therapist applied IASTM strokes for 20 seconds parallel to muscle fibers, followed by strokes for 20 seconds perpendicular to muscle fibers with the tool held at a 45° to the skin Treatment time was 3 minutes. Cryotherapy was applied for 10 minutes after the session. The treatment regimen will span over 3 weeks with a follow up frequency of 2 sessions per week.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization

INTERVENTIONS:
Other: Active Release Technique — active TrP was identified, and sustained and constant pressure was applied .for stretching of the SCM muscle, the patient performed contralateral lateral flexion and ipsilateral rotation of the head to achieve stretching, for trapezius the therapist performed lateral flexion of the neck.
  Arms: Active Release Technique
Other: Instrument Assisted Soft Tissue Mobilization — The therapist applied IASTM strokes for 20 seconds parallel to muscle fibers, followed by strokes for 20 seconds perpendicular to muscle fibers with the tool held at a 45° to the skin. .
  Arms: Instrument Assisted Soft Tissue Mobilization

SUMMARY:
Rationale of this research is to evaluate the outcome of active release technique and Instrument assisted soft tissue mobilization on trigger points in subjects with Migraine. The significance of this study is to identify which technique is superior in alleviating the symptoms of migraine. This study will help gather evidence on the practice of incorporating trigger point therapy in the treatment of Migraine.

DETAILED DESCRIPTION:
Migraine is a neurological condition that typically causes painful headache attacks lasting from four to 72 hours that occur with additional symptoms, such as sensitivity to light, sound, smell, or touch. Migraines occur most frequently in the morning, especially upon waking. Migraines can be triggered by stress or hormones. Migraine attacks are debilitating and can hinder the day to day activities and productivity of the patient. The purpose of the study was to evaluate the effects of active release technique and instrument assisted soft tissue mobilization on trigger points. It was a randomized, controlled trial, conducted among migraine patients. Sample size was 54 by using Epitool software. Participants were randomly assigned to the intervention or control group after a baseline assessment with a lottery ticket and an opaque envelope.All participants in both groups were evaluated on baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Both male and female 18-30 years Trigger points in Trapezius , Sternocleidomastoid and Sub-occipitals (Identified using Travel and Simmons Criteria) Migraine without Aura Subjects were cognitively capable and competent to follow the instructions

Exclusion Criteria:

Dysfunctions in the temporomandibular joint. Participant with a history of basilar migraine or hemiplegic migraine Fracture of Cervical Spine Currently on Medication for Migraine

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rate Scale: | 3rd week
  Numeric Pain Rate Scale used to measure pain intensity.
Cervical Goniometer | 3rd week
  Cervical Goniometer used to assess cervical ranges.

SECONDARY OUTCOMES:
HIT-6 Headache Impact Test | 3rd week
  The Headache Impact Test (HIT) is a tool used to measure the impact headaches have on your ability to function on the job, at school, at home and in social situations.

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Gulberg green campus of Riphah International University, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burch RC, Loder S, Loder E, Smitherman TA. The prevalence and burden of migraine and severe headache in the United States: updated statistics from government health surveillance studies. Headache. 2015 Jan;55(1):21-34. doi: 10.1111/head.12482. Erratum In: Headache. 2015 Feb;55(2):356. PMID 25600719
- [Background] Amiri P, Kazeminasab S, Nejadghaderi SA, Mohammadinasab R, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Migraine: A Review on Its History, Global Epidemiology, Risk Factors, and Comorbidities. Front Neurol. 2022 Feb 23;12:800605. doi: 10.3389/fneur.2021.800605. eCollection 2021. PMID 35281991
- [Background] Garcia-Leiva JM, Hidalgo J, Rico-Villademoros F, Moreno V, Calandre EP. Effectiveness of ropivacaine trigger points inactivation in the prophylactic management of patients with severe migraine. Pain Med. 2007 Jan-Feb;8(1):65-70. doi: 10.1111/j.1526-4637.2007.00251.x. PMID 17244105